CLINICAL TRIAL: NCT04756089
Title: Breast Stimulation for Labor Induction: a Parallel-group Randomized Controlled External Pilot Study of Acceptability and Feasibility
Brief Title: Stimulation Therapy for Inducing Mothers
Acronym: STIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2000029909
Record Dates: First submitted 2021-02-10; First posted 2021-02-16 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Induced; Birth; Labor Long; Labor Pain; Breast Pumping; Lactation Induced
MeSH Terms: conditions — Labor Pain; Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: This is a pilot feasibility and acceptability study of a randomized clinical trial of pregnant women at 36 weeks of gestation and greater randomized to one of two arms at Yale New Haven Hospital: (1) breast stimulation by hand or with a breast pump versus (2) exogenous intravenous oxytocin infusion (standard of care, control). The pilot study will be randomized since one of the goals is to evaluate whether the idea of randomization would be acceptable to patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast stimulation (Experimental): Participants randomized to the breast stimulation will use breast stimulation by hand or with an electronic breast pump (intervention) to stimulate labor.
  Interventions: Device: Electronic breast pump
- Exogenous oxytocin intravenous infusion (Active Comparator): Participants randomized to the standard care arm will use exogenous oxytocin intravenous infusion to stimulate labor.
  Interventions: Other: Exogenous oxytocin intravenous infusion

INTERVENTIONS:
Device: Electronic breast pump — Participants randomized to the breast stimulation will use breast stimulation by hand or with an electronic breast pump (intervention) to stimulate labor.
  Other Names: Medela Symphony pump
  Arms: Breast stimulation
Other: Exogenous oxytocin intravenous infusion — Participants randomized to the standard care arm will use exogenous oxytocin intravenous infusion to stimulate labor.
  Arms: Exogenous oxytocin intravenous infusion

SUMMARY:
This is a pilot feasibility and acceptability study of a randomized clinical trial of pregnant women at 36 weeks of gestation and greater randomized to one of two arms at Yale New Haven Hospital: (1) Breast stimulation by hand or with an electronic breast pump (intervention) compared to (2) Exogenous oxytocin intravenous infusion (current standard of care, control). The pilot study will be randomized since one of the goals is to evaluate whether the idea of randomization would be acceptable to patients.

DETAILED DESCRIPTION:
Almost four million women give birth each year in the United States with more than 27% of them undergoing induction of labor. Generally, labor induction is indicated when the benefits of expeditious delivery outweigh the risks of continuing the pregnancy. Additionally, labor induction is increasingly seen as a potentially therapeutic intervention even in the absence of any pregnancy complication for nulliparas after 39 weeks of gestation. However, induction of labor is usually associated with a longer latent phase compared to spontaneous labor, and may result in the need for cesarean delivery at an individual level when an induction attempt fails. Furthermore, it has been shown that women who are induced are less likely to be satisfied with their birth experience compared to those with spontaneous labor. Women are increasingly interested in a less medicalized birth experience and desire more control during their labor process. Lastly, the cost and infrastructure that would be required to universally apply routine induction of labor at 39 weeks of gestation are frequently cited as prohibitive, despite its associated improved outcomes.

Breast stimulation has been purported as a natural and inexpensive non-medical method for inducing labor that may give patients greater control over the process and have other potential clinical benefits. It is thought that breast stimulation induces uterine contractility by increasing the level of endogenous oxytocin hormone. Breast stimulation was historically used successfully for inducing contractions for the purposes of contraction stress testing.

A Cochrane review was performed in 2010 that compared breast stimulation with either no intervention or oxytocin infusion for labor induction. They found a significant reduction in the number of women not in labor at 72 hours (62.7% vs. 93.6%, RR 0.67, 95% CI 0.60-0.74) and the incidence of postpartum hemorrhage (0.7% vs. 6%, RR 0.16, 95% CI 0.03-0.87) among those who underwent breast stimulation compared to those who did not receive any intervention for induction. There were no benefits seen when comparing women who underwent breast stimulation versus those who received oxytocin alone. Despite the promising findings, the Cochrane Review raised the possibility of safety concerns due to one trial that reported four perinatal deaths (three in the breast stimulation group and one in the oxytocin group). However, that study was conducted in India, women were not monitored during breast stimulation, there was no clearly reported method of randomization, and there were very few study details divulged. The Cochrane Review ultimately had limited conclusions for several reasons. First, most included studies compared breast stimulation to no intervention, which is not the appropriate alternative when it has been determined that a labor induction is indicated. Additionally, most studies involved breast stimulation by hand at home for 1-3 hours per day and included only women with "low-risk" or un-specified risk pregnancies.

Only one previous trial has tested breast stimulation by breast pump, which showed that the time to reach the active phase of labor was significantly reduced among women who underwent breast stimulation compared to those who received oxytocin in the hospital setting. There was no difference in the length of labor between groups once women were considered to be in the active phase of labor or mode of delivery, but the trial included just 62 women. Reassuringly, only one of the 30 women assigned to breast stimulation requested discontinuation due to nipple soreness after 5.5 hours of intermittent stimulation.

Breast stimulation by hand or with an electronic breast pump is a biologically plausible method of labor induction that can potentially allow labor induction to be more efficient and may also have other benefits. These may include effects related to improved uterine contractility (e.g., successful labor induction and decreased postpartum hemorrhage risk), patient satisfaction with the induction process, and the stimulation of endogenous oxytocin which may improve postpartum breastfeeding and positive emotional responses. A well-designed randomized clinical trial is needed to evaluate the efficacy and safety of breast stimulation, particularly in comparison to the clinical alternative (use of exogenous oxytocin).

This is a proposed prospective parallel group randomized controlled external pilot study of breast stimulation by hand or with an electronic breast pump compared to exogenous oxytocin infusion to assess acceptability and feasibility prior to conducting a large non-inferiority randomized trial.

The two arms in this study are: (1) Breast stimulation by hand or with an electronic breast pump (intervention) compared to (2) Exogenous oxytocin intravenous infusion (current standard of care, control).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Age 18 years and older
4. Gestational age 36 weeks and greater at randomization
5. Vertex-presenting singleton gestation, or presenting gestation (a.k.a. Fetus A) is vertex-presenting in a multiple gestation
6. Undergoing induction of labor
7. Planned to undergo initiation of exogenous oxytocin infusion by their maternity care provider
8. Absence of tachysystole (defined as more than 5 contractions in 10 minutes averaged over 30 minutes), recurrent variable or late fetal decelerations, and bradycardia in the prior 30 minutes before randomization

Exclusion Criteria:

1. Unable to understand English
2. Planned for cesarean delivery or contraindication to labor by institutional policy (e.g., placenta previa, vasa previa, active genital herpes infection, uncontrolled HIV infection, previous transmural myomectomy)
3. Fetal demise
4. Major fetal anomaly suspected prenatally (defined as a fetal anomaly with anticipated neonatal intensive care unit admission)
5. Suspected fetal growth restriction (EFW <10th percentile)
6. Suspected alloimmunization
7. Unexplained active vaginal bleeding
8. History of mastectomy, breast lumpectomy, or contraindication to use of electronic breast pump
9. Known allergic reactions to components of the electronic breast pump or to synthetic oxytocin intravenous solution
10. Impairment of upper extremity motor function (e.g., quadriplegia)
11. Significantly impaired consciousness or executive function (e.g., intubated or sedated)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-03-13 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Recruitment (enrollment) rate | 3 months
  Determine the rate of eligible women who consent and enroll in the study among eligible women who are approached by research study staff.
Adherence rate | 3 months
  Determine the rate of randomized women who remain in the trial and complete all study procedures as outlined in the protocol among all women who are consented and randomized to study intervention.
Cross-over frequencies | 3 months
  Determine the percentage of women in each study intervention arm who cross over to the other study arm (i.e. cross-over from breast stimulation to exogenous intravenous oxytocin infusion in less than 2 hours, or cross-over from exogenous intravenous oxytocin infusion to breast stimulation) prior to their delivery

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stark EL, Athens ZG, Son M. Intrapartum nipple stimulation therapy for labor induction: a randomized controlled external pilot study of acceptability and feasibility. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100575. doi: 10.1016/j.ajogmf.2022.100575. Epub 2022 Jan 15. PMID 35042047